CLINICAL TRIAL: NCT04963153
Title: Phase Ib Trial of Erdafitinib Combined With Enfortumab Vedotin Following Prior Therapies for Metastatic Urothelial Carcinoma With FGFR2/3 Genetic Alterations.
Brief Title: Testing Combination Erdafitinib and Enfortumab Vedotin in Metastatic Bladder Cancer After Treatment With Chemotherapy and Immunotherapy
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2021-07069; NCI-2021-07069 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MCC 21460; 10483 (Other: Ohio State University Comprehensive Cancer Center LAO); 10483 (Other: CTEP); UM1CA186644 (NIH)
Record Dates: First submitted 2021-07-14; First posted 2021-07-15 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-10

CONDITIONS: Locally Advanced Bladder Urothelial Carcinoma; Locally Advanced Renal Pelvis Urothelial Carcinoma; Locally Advanced Ureter Urothelial Carcinoma; Locally Advanced Urethral Urothelial Carcinoma; Locally Advanced Urothelial Carcinoma; Metastatic Bladder Urothelial Carcinoma; Metastatic Renal Pelvis Urothelial Carcinoma; Metastatic Ureter Urothelial Carcinoma; Metastatic Urethral Urothelial Carcinoma; Metastatic Urothelial Carcinoma; Recurrent Bladder Urothelial Carcinoma; Recurrent Renal Pelvis Urothelial Carcinoma; Recurrent Ureter Urothelial Carcinoma; Recurrent Urethral Urothelial Carcinoma; Recurrent Urothelial Carcinoma; Stage IIIB Bladder Cancer AJCC v8; Stage IV Bladder Cancer AJCC v8; Stage IV Renal Pelvis Cancer AJCC v8; Stage IV Ureter Cancer AJCC v8; Stage IV Urethral Cancer AJCC v8
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Ureteral Neoplasms; Urethral Neoplasms | interventions — Specimen Handling; enfortumab vedotin; erdafitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (erdafitinib, enfortumab vedotin) (Experimental): Patients receive erdafitinib PO QD on days 1-28 of each cycle and enfortumab vedotin IV over 30 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo CT and blood sample collection throughout the trial and may undergo echocardiography or MUGA scan during screening and bone scan throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Echocardiography Test; Drug: Enfortumab Vedotin; Drug: Erdafitinib; Procedure: Multigated Acquisition Scan

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo echocardiography
  Other Names: EC; Echocardiography
Drug: Enfortumab Vedotin — Given IV
  Other Names: AGS 22ME; AGS-22M6E; Anti-Nectin 4 ADC ASG-22CE; Anti-nectin-4 Monoclonal Antibody-Drug Conjugate AGS-22M6E; ASG 22CE; ASG-22CE; ASG22CE; Enfortumab Vedotin-ejfv; Padcev
Drug: Erdafitinib — Given PO
  Other Names: Balversa; JNJ 42756493; JNJ-42756493; JNJ42756493
Procedure: Multigated Acquisition Scan — Undergo MUGA scan
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; Gated Heart Pool Scan; MUGA; MUGA Scan; Multi-Gated Acquisition Scan; Radionuclide Ventriculogram Scan; Radionuclide Ventriculography; RNV Scan; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning

SUMMARY:
This phase Ib trial evaluates the best dose, potential benefits, and/or side effects of erdafitinib in combination with enfortumab vedotin in treating patients with bladder cancer that has spread from where it first started (primary site) to other places in the body (metastatic) and possesses genetic alterations in FGFR2/3 genes. Erdafitinib is in a class of medications called kinase inhibitors. It works by blocking the action of an abnormal FGFR protein that signals cancer cells to multiply. This may help keep cancer cells from growing and may kill them. Enfortumab vedotin is a monoclonal antibody, enfortumab, linked to an anticancer drug called vedotin. It works by helping the immune system to slow or stop the growth of cancer cells. Enfortumab attaches to a protein called nectin-4 on cancer cells in a targeted way and delivers vedotin to kill them. It is a type of antibody-drug conjugate. Giving erdafitinib in combination with enfortumab vedotin may shrink or stabilize metastatic bladder cancer with alterations in FGFR 2/3 genes.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility and safety of erdafitinib when combined with enfortumab vedotin (EV) for patients with metastatic urothelial carcinoma (mUC) harboring FGFR2/3 activating genomic alterations who are progressing following platinum-based chemotherapy and PD1/L1 inhibitors.

II. To determine the maximally tolerated dose (MTD) and the recommended phase 2 dose (RP2D) of EV when combined with erdafitinib.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To observe and record overall response rate (ORR). III. To observe and record duration of response (DOR). IV. To observe and record progression-free survival (PFS). V. To observe and record overall survival (OS).

EXPLORATORY OBJECTIVES:

I. Assess association of tumor PD-L1, nectin-4 protein, FGFR3, cell lineage markers and progression markers expression with response.

II. Use commercial tissue/plasma next generation sequencing (NGS) assay to confirm FGFR status as well as to describe the genomic landscape of metastatic UC.

III. Use commercial liquid NGS assay to assess genomic changes by circulating tumor (ct)-deoxyribonucleic acid (DNA) assessment to study mechanisms of resistance with treatment.

IV. Assess pharmacokinetic (PK) of monomethyl auristatin E (MMAE) and erdafitinib.

OUTLINE: This is a dose-escalation study of enfortumab vedotin in combination with fixed dose erdafitinib followed by a dose-expansion study of the drug combination.

Patients receive erdafitinib orally (PO) once daily (QD) on days 1-28 of each cycle and enfortumab vedotin intravenously (IV) over 30 minutes on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity. Patients also undergo computed tomography (CT) and blood sample collection throughout the trial and may undergo echocardiography or multigated acquisition (MUGA) scan during screening and bone scan throughout the study.

After completion of study treatment, patients are followed up every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically documented locally advanced (T4b, any N; or any T, N 2-3) or metastatic (M1, Stage IV; or metastatic recurrence after locoregional treatment) urothelial carcinoma (including renal pelvis, ureters, urinary bladder, urethra). Patients with mixed histologies are required to have a dominant transitional cell pattern
* Patients who had disease progression during or following treatment with at least one platinum-containing regimen (e.g., gemcitabine and cisplatin [GC], methotrexate, vinblastine, doxorubicin and cisplatin [MVAC], carboplatin and gemcitabine [Carbo-Gem]) and an immune checkpoint inhibitor (PD-1/ PD-L1 inhibitor including but not limited to: atezolizumab, pembrolizumab, durvalumab, avelumab, and nivolumab)

  * Received a first-line platinum-containing regimen in the metastatic setting or for inoperable locally advanced disease
  * Or received neo/adjuvant platinum-containing therapy for localized muscle-invasive UC, with recurrence/progression =< 12 months following completion of therapy
  * Patients who received immune checkpoint inhibitor therapy in the neoadjuvant/adjuvant setting and had recurrent or progressive disease either during therapy or within 12 months of therapy completion are eligible. This criterion does not apply if the checkpoint inhibitor is contraindicated
* Patients with metastatic urothelial carcinoma who are cisplatin-ineligible and progressed on upfront immune checkpoint inhibitor; or ineligible/refused immune checkpoint inhibitor therapy will be eligible for this trial
* Patient who received prior antibody drug conjugate such as sacituzumab govitecan are allowed
* Patients must have measurable disease, as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. Previously irradiated lesions cannot be counted as target lesions unless there has been demonstrated progression in the lesion since radiotherapy and no other lesions are available for selection as target lesions
* Patients must have FGFR2/3 activating alterations identified by tumor tissue or plasma ctDNA profiling using a Clinical Laboratory Improvement Act (CLIA) certified College of American Pathologists (CAP) accredited platform
* Age >= 18 years, for ability to comply with protocol

  * Because no dosing or adverse event data are currently available on the use of erdafitinib in combination with enfortumab vedotin in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Absolute neutrophil count >= 1,500/mcL (within 14 days prior to beginning trial treatment)
* Platelets >= 100,000/mcL (within 14 days prior to beginning trial treatment)
* Hemoglobin >= 9 g/dL (within 14 days prior to beginning trial treatment)
* Measured or calculated creatine clearance (CrCl) >= 30 ml/min (glomerular filtration rate [GFR] can also be used in place of creatinine CrCl) (within 14 days prior to beginning trial treatment)
* Total bilirubin =< 1.5 x ULN (institutional upper limit of normal) OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 x ULN (within 14 days prior to beginning trial treatment)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 2.5 x institutional ULN (=< 5 x ULN for subjects with liver metastasis) (within 14 days prior to beginning trial treatment)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression (CNS metastases have been clinically stable for at least 4 weeks prior to screening and baseline scans show no evidence of new or enlarged metastasis)
* Patients with a history of prostate cancer (T2NXMX or lower with Gleason score =< 7) treated with definitive intent (surgically or with radiation therapy) at least 1 year prior to study entry are eligible, provided that the subject is considered prostate cancer-free and the following criteria are met:

  * Patients who have undergone radical prostatectomy must have undetectable prostate specific antigen (PSA) for > 1 year and at screening
  * Patients who have had radiation must have a PSA doubling time > 1 year (based on at least 3 values determined >1 month apart) and a total PSA value that does not meet Phoenix criteria for biochemical recurrence (i.e., < 2.0 ng/mL above nadir)
  * Patients with untreated low-risk prostate cancer (Gleason score =< 6) on active surveillance with PSA doubling time >1 year (based on at least 3 values determined > 1 month apart) are also eligible
* Patients who have undergone an ophthalmologic examination and have no active eye disease which would be likely to increase the risk of eye toxicity
* The effects of erdafitinib and enfortumab vedotin on the developing human fetus are unknown. For this reason and because FGFR inhibitors and humanized antibody-drug conjugate (ADC) agents are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and 3 months after completion of erdafitinib and enfortumab vedotin administration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 5 months after completion of erdafitinib and enfortumab vedotin administration
* Ability to understand and willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy, targeted therapies, immunotherapy, or treatment with an investigational anticancer agent within 2 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (including ongoing sensory or motor neuropathy of grade 2 or higher) (i.e., have residual toxicities > grade 1 or returned to baseline) with the exception of alopecia. Subjects with =< grade 2 immunotherapy- related hypothyroidism or panhypopituitarism may be enrolled when well-maintained/controlled on a stable dose of hormone replacement therapy (if indicated). Subjects with ongoing >= grade 3 immunotherapy-related hypothyroidism or panhypopituitarism are excluded. Subjects with ongoing immunotherapy related colitis, uveitis, myocarditis, or pneumonitis or subjects with other immunotherapy related adverse events (AEs) requiring high doses of steroids (> 20 mg/day of prednisone or equivalent) are excluded
* Patients who have previously received enfortumab vedotin or other MMAE-based ADCs
* Patients who have had prior treatment with an FGFR inhibitor
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to erdafitinib and enfortumab vedotin
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with a history of any corneal or retinal abnormality likely to increase the risk of eye toxicity
* Patients with uncontrolled intercurrent illness and currently receiving systemic antimicrobial treatment for active infection (viral, bacterial, or fungal) at the time of starting treatment. Routine antimicrobial prophylaxis is permitted
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Subjects who have received radiotherapy within 2 weeks prior to start of treatment. Subject must have recovered adequately from the toxicity from the intervention prior to starting study treatment
* Patients with uncontrolled diabetes. Uncontrolled diabetes is defined as hemoglobin A1c (HbA1c) >= 8% or HbA1c 7% to < 8% with associated diabetes symptoms (polyuria or polydipsia) that are not otherwise explained
* Subjects who have received major surgery within 4 weeks prior to start of treatment. Subject must have recovered adequately from complications from the intervention prior to starting study treatment
* Subjects who have received a prior allogeneic stem cell or solid organ transplant
* Has persistent phosphate level > ULN during screening (within 14 days of treatment and prior to cycle 1 day 1) and despite medical management
* Has a history of or current uncontrolled cardiovascular disease including:

  * Unstable angina, myocardial infarction, or known congestive heart failure class II-IV within the preceding 12 months; cerebrovascular accident or transient ischemic attack within the preceding 3 months
  * Any of the following: sustained ventricular tachycardia, ventricular fibrillation, Torsades de Pointes, cardiac arrest, Mobitz II second degree heart block or third degree heart block; known presence of dilated, hypertrophic, or restrictive cardiomyopathy
  * Corrected QT interval (QTc) prolongation as confirmed by triplicate assessment at screening (Fridericia;QTc > 480 milliseconds)
* Subjects with a history of another invasive malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy. Subjects with nonmelanoma skin cancer or carcinoma in situ of any type (if complete resection was performed) are allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-07-07 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 2 years
Recommended phase II dose | Up to 28 days
Maximum tolerated dose of enfortumab vedotin | Up to 28 days
  The highest dose of enfortumab vedotin in combination with fixed dose erdafitinib that does not cause unacceptable side effect.

SECONDARY OUTCOMES:
Overall response rate | Up to 2 years from study enrollment
  Will be summarized using descriptive statistics including two-sided 95% confidence interval (CI) based on Clopper-Pearson method.
Duration of response | Time from complete response or partial response (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years from study enrollment
  Will be summarized using mean, standard deviation, median, and range.
Progression free survival | Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years
  Kaplan-Meier curve estimates of medians and their corresponding 95% CIs will be calculated.
Overall survival | Up to 2 years from study enrollment
  Kaplan-Meier curve estimates of medians and their corresponding 95% CIs will be calculated.

OTHER OUTCOMES:
PD-L1, Nectin-4, FGFR3/phosphor-FGFR3, cell lineage and progression marker expression | Up to 2 years from study enrollment
Tumor subtyping, tumor microenvironment, and mutations associated with treatment response | Up to 2 years from study enrollment
  Will be evaluated based on pre-treatment sequencing data.
Mechanisms of resistance and response | Up to 2 years from study enrollment
  Will be evaluated through peripheral blood circulating tumor deoxyribonucleic acid (DNA). Methods of analysis may include but not limited to, immunohistochemistry, next-generation sequencing of DNA and ribonucleic acid, and immunoassays.
Pharmacokinetics (PK) | Up to 2 years from study enrollment
  PK analysis will be performed to explore the relationship between drug exposure, toxicity and response.

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Jain, Principal Investigator — University Health Network Princess Margaret Cancer Center LAO
Locations (10):
- United States (9):
  - Los Angeles General Medical Center, Los Angeles, California
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - NYP/Weill Cornell Medical Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
- University Health Network-Princess Margaret Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2025-02-06): https://cdn.clinicaltrials.gov/large-docs/53/NCT04963153/ICF_000.pdf